CLINICAL TRIAL: NCT03995290
Title: The Use of Patient-Specific 3D Printed Anatomic Models in Pre-Operative Planning and Patient Engagement to Improve Hip Arthroscopy Outcomes
Brief Title: 3D Modeling to Improve Hip Arthroscopy Outcomes
Status: Terminated | Type: Observational
Why Stopped: Loss of funding.
Sponsor: The Hawkins Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00086834
Record Dates: First submitted 2019-06-18; First posted 2019-06-24 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 3D Hip Model from Pre-operative CT scan — A printed 3D model will be created based off of the patient's standard of care preoperative CT scan.

SUMMARY:
This study will pilot the use of 3D printed models of the hip, for use in pre-operative planning and patient communication to improve clinical outcomes and patient engagement. This method will be implemented in the setting of femoroacetabular impingement (FAI), with the goal of identifying and measuring specific anatomical pathologies and impingement (range of motion) risks, to communicate a pre-operative plan to both the surgical team, and the patient.

DETAILED DESCRIPTION:
Following a standard of care pre-operative CT scan, a 3D rendering of the CT scan will be completed. The de-identified CT Scan data will be transferred to the Clemson University Bioengineering Department, and a 3D modeling software will convert it to a computer model that will then be 3D printed. During the doctor-patient pre-operative consultation, the 3D Printed model will be used to assist the doctor in describing the patient's pathology and upcoming surgical procedure. In this pilot study, the surgeon will make measurements and estimates of resection for the femoroplasty and acetabuloplasty off of 2D CT scan, MRI, and x-rays. This will then be compared quantitatively to the results of the 3D model/3D printing measurements. Surgeon debriefings will occur postoperatively to determine the benefit of the model and how well it matched up to what the surgeon experienced during the surgery.

FAI involves complex anatomic morphology which can be unique to each patient. A thorough understanding of the type and specifically location of impingement is paramount to successful results if surgery is required. 2D imaging has limitations when analyzing a 3D anatomic lesion. 3D printed hip models have the potential to provide superior preoperative planning and subsequent surgical results. In addition, 3D models can potentially improve patient understanding, expectations, and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Surgical candidate for a hip arthroscopy for the treatment of femoroacetabular impingement
* Subject is willing to sign the informed consent.
* Subject is at least 18 years of age.

Exclusion Criteria (n/a)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject will be approached for participation in this study after the subject has made the decision to undergo a hip arthroscopy procedure and will be receiving a standard of care hip CT Scan. Patients who meet all criteria will be offered enrollment into the study.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Resection Measurement Variations | Pre-operative through date of surgery: Resection measurements will be collected intra-operatively and compared to the pre-operative estimations.
  The surgeon will make estimates of resection for the femoroplasty and acetabuloplasty based on standard pre-operative imaging (in millimeters). The surgeon will also make estimates based on the 3D model/3D printing measurements. Actual resection measurements will be collected intra-operatively and compared to the surgeon's pre-operative predictions based on the 3D model and the standard imaging techniques (in millimeters).

CONTACTS AND LOCATIONS:
Locations (1):
- Steadman Hawkins Clinic of the Carolinas - Greenville Health System, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No